CLINICAL TRIAL: NCT00004648
Title: Studies of Hereditary Hemorrhagic Telangiectasia: Screening Methods for Pulmonary Arteriovenous Malformations; Prevalence of Pulmonary and Cerebral Arteriovenous Malformations; Prevalence of Cardiac Valve Abnormalities; and Identification of Modifier Genes
Brief Title: Studies of Hereditary Hemorrhagic Telangiectasia
Status: Completed | Type: Observational
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: University of Vermont (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Other Study IDs: 199/11711; UVT-651
Record Dates: First submitted 2000-02-24; First posted 2000-02-25 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2001-12

CONDITIONS: Telangiectasia, Hereditary Hemorrhagic
Keywords: genetic diseases and dysmorphic syndromes; hematologic disorders; hereditary hemorrhagic telangiectasia; rare disease; Osler-Rendu-Weber disease
MeSH Terms: conditions — Telangiectasia, Hereditary Hemorrhagic; Genetic Diseases, Inborn; Hematologic Diseases; Rare Diseases

SUMMARY:
OBJECTIVES: I. Examine screening modalities for pulmonary vascular arteriovenous malformation (PAVM) in individuals with endoglin mutations.

II. Examine the prevalence of cerebral arteriovenous malformations (CAVM) in individuals with hereditary hemorrhagic telangiectasia (HHT).

III. Investigate whether modifier genes exist that determine which individuals with HHT due to an endoglin mutation develop PAVMs and which develop CAVMs.

IV. Investigate the frequency of cardiac valve abnormalities in individuals affected with HHT due to an endoglin mutations.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: Patients with hereditary hemorrhagic telangiectasia (HHT) undergo 5 different screening methods to determine which method is most effective in detecting arteriovenous malformations (AVM). Patients may participate in more than one screening method.

In part 1, patients undergo 3 different screening techniques (e.g., pulse oximetry, spiral computed tomography (CT), and contrast echocardiography) to detect pulmonary arteriovenous malformations (PAVM).

Patients in part 2 undergo magnetic resonance imaging (MRI) using gadolinium as the contrasting agent for AVM in the brain, known as cerebral arteriovenous malformations (CAVM). For pregnant women, this procedure may only take place if there is clinical evidence that suggests CAVM.

In part 3, Doppler ultrasound is used to screen for hepatic arteriovenous malformations (HAVM). The abdomen of each patient is viewed to detect AVM in the liver.

Patients in part 4 undergo echocardiograms as the screening method used to determine common heart valve abnormalities.

In part 5, blood samples are drawn from patients and analyzed to locate modifier genes as a possibility in determining severity of HHT.

ELIGIBILITY:
* Osler-Rendu-Weber disease (or hereditary hemorrhagic telangiectasia)

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 65
Dates: Start 1996-05

CONTACTS AND LOCATIONS:
Overall Officials: Alan Guttmacher, Study Chair — University of Vermont